CLINICAL TRIAL: NCT01549106
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and the Effect of Food and Ketoconazole on the Pharmacokinetics of IPI-145 When Administered to Healthy Adult Subjects
Brief Title: IPI-145 Single Ascending, Multiple Ascending, Food Effect and Drug-Drug-Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IPI-145-01; 2011-001944-31 (EudraCT Number)
Record Dates: First submitted 2012-02-10; First posted 2012-03-08 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — duvelisib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPI-145 (Experimental)
  Interventions: Drug: IPI-145
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IPI-145 — Single ascending dose up to 6 cohorts; multiple ascending dose up to 4 cohorts; food effect arm; ketoconazole drug interaction study
  Arms: IPI-145
Drug: Placebo — Single ascending dose up to 6 cohorts; multiple ascending dose up to 4 cohorts; food effect arm
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of IPI-145 after single and repeat oral administration, and to evaluate the effects of food and ketoconazole on the plasma pharmacokinetics of IPI-145.

ELIGIBILITY:
Inclusion Criteria:

1. Gender : male or female
2. Age : 18-55 years, inclusive
3. Body Mass Index (BMI) : 18.0-30.0 kg/m2
4. Medical history without major pathology
5. For males only: Willingness to use adequate contraception from the time of dosing and not donate sperm until 3 months after the follow-up visit
6. Females who have a negative pregnancy test at screening and on each admission, and are of non-childbearing potential. Females of non-childbearing potential are defined as women who are surgically sterile or post-menopausal (defined as at least 1 year post cessation of menses and follicular stimulating hormone (FSH) >23.0 mIU/mL)
7. Willing and able to sign the written Informed Consent Form (ICF)

Exclusion Criteria:

1. Previous participation in the current study
2. Evidence of clinically relevant pathology
3. History of relevant drug and/or food allergies
4. Part 4 only: Known or suspected adverse reaction or contraindication to the imidazole class of drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessments consisting of adverse events, vital signs, 12-lead ECG, clinical laboratory tests and physical examinations will be performed following IPI-145 single and repeat oral administration in healthy subjects | 8 months
Plasma concentrations of IPI-145 and metabolites | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (1):
- PRA International, Zuidlaren, Netherlands